CLINICAL TRIAL: NCT02962479
Title: Is the Human Microbiome Altered in Patients With Axial Spondyloarthritis?
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Eyal Kedar (Other)
Responsible Party: Sponsor-Investigator, Eyal Kedar, Rheumatologist, St. Lawrence Health System
Organization: St. Lawrence Health System (Other)
Other Study IDs: EK001
Record Dates: First submitted 2016-11-08; First posted 2016-11-11 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Axial Spondyloarthritis; Ankylosing Spondylitis
MeSH Terms: conditions — Axial Spondyloarthritis; Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Subjects will have the option to provide additional consent for specimens to be retained by the research team indefinitely for research purposes. These samples will be identified only by the numeric study ID; no personally identifying information will be associated with the retained samples. The samples could be used to make new products, tests or findings, which may have value and may be developed and owned by the research team and/or others. Investigators will not be able to provide subjects with results from any future research that is done using their samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- TNF blocker-naïve ankylosing spondylitis patients
- TNF blocker-exposed ankylosing spondylitis patients
- TNF blocker-naïve nrSpA patients
- TNF blocker-exposed nrSpA patients
- Healthy Participants

SUMMARY:
This study aims to compare biological communities in stool samples obtained from age, diet and BMI-matched subjects in five study groups: subjects with ankylosing spondylitis (AS) never treated with tumor necrosing factor (TNF) inhibitors, subjects with ankylosing spondylitis previously or currently treated with TNF inhibitors, subjects with non-radiographic axial spondyloarthritis (nrSpA) never treated with tumor necrosing factor (TNF) inhibitors, subjects with non-radiographic axial spondyloarthritis previously or currently treated with TNF inhibitors and healthy participants.

The differences in fecal microbiota composition will be explored using shotgun metagenomic sequencing through the University of Washington. The investigators predict that this study will confirm a significant difference between the fecal microbiota composition (FMC) of both AS and nrSpA patients and controls.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Male or Female patients ≥18 years of age
* Additional Inclusion Criteria based on cohort

Exclusion Criteria:

* Current use of any pain-relieving medications other than NSAIDs, APAP and/or opioids
* Corticosteroid therapy or probiotic exposure within the last two weeks
* Antibiotic exposure within the past two months
* History of psoriasis or inflammatory bowel disease or reactive arthritis or any other chronic rheumatologic disease
* Active infection
* History of hepatitis B or C or HIV
* Active cancer or history of colon cancer or any form of chemotherapy or radiation within the past year
* Celiac disease
* Use of proton pump inhibitors within the prior two months
* History of clostridium difficile
* Pregnancy
* Active diarrhea (defined as a decrease in fecal consistency lasting four or more weeks)
* Additional Exclusion Criteria based on cohort

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: At least 50 subjects, male and female, aged 18 or older, will be recruited to the study and assigned to one of five groups:
  1. Ten TNF blocker-naïve ankylosing spondylitis patients
  2. Ten TNF blocker-exposed ankylosing spondylitis patients
  3. Ten TNF blocker-naïve nrSpA patietns
  4. Ten TNF blocker-exposed nrSpA patients
  5. Ten healthy age, diet and BMI-matched controls Inclusion and exclusion criteria will vary by study group. It is anticipated that the TNF-blocker naïve groups will be the most difficult to recruit, so these groups will serve as the baseline for age and diet matching for the other two groups. Up to seventy (70) additional TNF-treated axial SpA and healthy subjects may be asked to complete the dietary questionnaire, but will not provide stool samples unless age, diet and BMI-matched with a TNF-blocker-naïve axial SpA subject.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Weighted and unweighted UniFrac distances between stool samples from the five study groups | Within 1 month of baseline visit

CONTACTS AND LOCATIONS:
Locations (1):
- St. Lawrence Health System, Potsdam, New York, United States